CLINICAL TRIAL: NCT04063176
Title: Prospective Outpatient Registry of Myocardial Infarction Patients
Acronym: PROFILE-MI
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: PROFILE-MI
Record Dates: First submitted 2019-08-15; First posted 2019-08-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction, registry
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators enrolled 160 patients who visited Moscow state outpatient clinic №9 (and its two branches) within six months after acute myocardial infarction. The enrollment lasted from 01.03.2014 to 01.07.2015. The observation period is five years. During the first year after enrollment in the study, patients had follow-up visits every two months, from second-year every six months. Analysis of the prescribed therapy and its changes was carried out by the cardiologist in the clinic for the entire observation period, taking into account the concomitant diseases /indications/contraindications. Endpoints (the death, repeated cardiovascular complications (AMI, stroke), emergency hospitalization due to worsening of the main cardiovascular disease, the appearance of clinically significant cardiac arrhythmias, invasive interventions) were defined during out-patient visits and telephone contact

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone AMI and applied no later than 6 months. after discharge from the hospital to the Moscow outpatient clinic № 9 from March 1, 2014, to December 31, 2015;
* availability of discharge summary with confirmed AMI;
* permanent residence on the territory of Moscow and the Moscow region;
* the signing of informed consent to the processing of personal data.

Exclusion Criteria:

* patients with the absence of discharge summary from the hospital with a proven history of AMI;
* visit the clinic in a period exceeding six months from the AMI;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have undergone AMI and applied no later than 6 months after discharge from the hospital to the outpatient clinic № 9 or its branches from March 1, 2014 to December 31, 2015;
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
time to death, recurrent cardiovascular events (AMI, stroke), emergency hospitalization, lifethreatening arrhythmias. | 01.03.2014 - through study completion, an average of 5 year
  According to the results of monitoring will be determined a combined endpoint: the death, recurrent cardiovascular events, emergency hospitalization, lifethreatening arrhythmias

SECONDARY OUTCOMES:
Total mortality | 01.03.2014 - through study completion, an average of 5 year
  Determination of total mortality for any reason of patients enrolled in the Registry

CONTACTS AND LOCATIONS:
Overall Officials: Martsevich Yu Sergey, MD, PhD, professor, Study Chair — National Research Center for Preventive Medicine; Natalia P Kutishenko, Principal Investigator — National Research Center for Preventive Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Martsevich S.Yu., Kutishenko N.P., Sichinava D.P., Kalaydzhian Е.P. Prospective outpatient registry of myocardial infarction patients (PROFILE-MI): study design and first results (in russian) Cardiovascular Therapy and Prevention, 2018; 17(1): 81-86 — http://dx.doi.org/10.15829/1728-8800-2018-1-81-86
- See also: Kutishenko N.P.,Kalaydzhyan E.P.,Sichinava D.P.,Evdakov V.A.,Martsevich S.Yu.OUTPATIENT REGISTRY OF PATIENTS WITH ACUTE MYOCARDIAL INFARCTION(PROFILE-IM):DATA ON PREHOSPITAL THERAPY IN COMPARISON WITH THE LIS-3 REGISTRY.(In Russ.)RPC.2018;14(1):88-93 — https://doi.org/10.20996/1819-6446-2018-14-1-88-93
- See also: Kutishenko N.P., Sichinava D.P.,Kalaydzhyan E.P.,Evdakov V.A.,Kasparova E.A.,Martsevich S.Yu.Effect of Previous Cardiovascular Diseases on Long-Term Outcomes of Acute Myocardial Infarction:Data of the Outpatient Registry"PROFILE-IM". RPС.2018;14(5):741-7 — https://doi.org/10.20996/1819-6446-2018-14-5-741-746
- See also: Martsevich S.Yu., Kutishenko N.P., Kalaydzhyan E.P., Sichinava D.P., Evdakov V.A. Assessment of the Adequacy of Drug Choice in Patients with Acute Myocardial Infarction According to the PROFILE-IM Registry. RPC. 2019;15(2):224-229.(In Russ.) — https://doi.org/10.20996/1819-6446-2019-15-2-224-229
- See also: Sichinava D.P., Kalaydzhyan E.P., Kutishenko N.P., Martsevich S.Yu. Outpatient Register of Patients with Acute Myocardial Infarction: Assessment of the Hypertension Impact on Long-term Prognosis.RPC.2019;15(5):706-712.(In Russ.) — https://doi.org/10.20996/1819-6446-2019-15-5-706-712
- See also: Martsevich S.Yu.,Kutishenko N.P.,Sichinava D.P.,Kalaydzhyan E.P. The Main Cardiovascular Complications and Mortality Rates During the First One and a Half Years after Acute Myocardial Infarction: Data from the Prospective Outpatient Registry PROFILE-IM. — https://doi.org/10.20996/1819-6446-2020-06-11
- See also: Kalaydzhyan E.P., Martsevich S.Yu., Kutishenko N.P., Sichinava D.P., Drapkina O.M. Untapped Possibilities of Antiischemic Therapy after Acute Myocardial Infarction: Data from the PROFILE-IM Register.RPC. 2020;16(3):432-438. (In Russ.) — https://doi.org/10.20996/1819-6446-2020-10-22
- See also: Kalaydzhyan E.P., Kutishenko N.P., Lukina Yu.V., Sichinava D.P., Martsevich S.Yu., Drapkina O.M. The Study of Adherence to Drug Therapy at the Stage of Outpatient Follow-up in Patients with Acute Myocardial Infarction (Data from the PROFIL-IM Registry). — https://doi.org/10.20996/1819-6446-2023-02-04